CLINICAL TRIAL: NCT01329263
Title: Smoking Topography and Harm Exposure in Menthol Cigarettes
Acronym: MQAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH); National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Andrew Strasser, Associate Professor Department of Psychiatry, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 812369; R01CA120594 (NIH); R01CA130961 (NIH); P30ES013508 (NIH); P50CA143187 (NIH)
Record Dates: First submitted 2011-04-01; First posted 2011-04-05 (Estimated); Results first posted 2014-12-15 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2014-12

CONDITIONS: Cigarette Smoking Toxicity
Keywords: menthol cigarettes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nonmenthol (Experimental): Participants switch from menthol to non-menthol cigarettes.
  Interventions: Other: Menthol to non-menthol
- Menthol (No Intervention): Participants smoke own brand of menthol cigarettes.

INTERVENTIONS:
Other: Menthol to non-menthol — Switch from smoking menthol to non-menthol cigarettes.
  Arms: Nonmenthol

SUMMARY:
This study will examine how menthol affects smoking when menthol smokers switch to non-menthol cigarettes. Participants will smoke their preferred brand (control) or Camel Crush cigarettes, which have the ability to be menthol or non-menthol. Participants given Camel Crush cigarettes will smoke them as menthol, then non-menthol cigarettes for 15 days each. Participants will provide breath and urine samples, track cigarette usage and complete smoking topography assessments of smoking behavior.

DETAILED DESCRIPTION:
This study will examine how menthol affects smoking behaviors and biomarker level when menthol smokers switch to non-menthol cigarettes. Participants will initially smoke their preferred brand (control) cigarettes, followed by smoking Camel Crush cigarettes, which have the ability to be menthol or non-menthol. Participants given Camel Crush cigarettes will smoke them as menthol, then non-menthol cigarettes for 15 days each. Participants will provide breath and urine samples to measure smoke exposures, track cigarette usage to establish changes in daily cigarette consumption and complete smoking topography assessments of smoking behavior, such as puff volume.

ELIGIBILITY:
Inclusion Criteria:

* Self-report smoking daily cigarettes
* Self-report smoking menthol flavored cigarettes
* Not currently trying to quit or planning to quit in the next 2 months.
* Interested in trying a novel cigarette product and willing to smoke a non-menthol cigarette
* Self-report smoking only filtered commercially made cigarettes

Exclusion Criteria:

* Self-report drinking equal to or greater than a certain number of alcohol-containing drinks per week
* Self report using any nicotine replacement products or nicotine-containing products other than cigarettes
* Self-report substance use disorders in the last 5 years
* Self-report current Axis I psychiatric disorders
* Self-report past history of Axis I psychiatric disorders other than depression
* Self-report myocardial infarction, angina or abnormal rhythms requiring medication
* Self-report use of select medications and illicit drugs within past six months
* Females must not be currently pregnant, planning a pregnancy during the study, or currently breastfeeding/lactating
* Provide a baseline carbon monoxide (CO) reading < 10 ppm at initial session
* Inability to provide informed consent or complete any of the study tasks as determined by the Principal Investigator

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2010-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew A Strasser, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Strasser AA, Ashare RL, Kaufman M, Tang KZ, Mesaros AC, Blair IA. The effect of menthol on cigarette smoking behaviors, biomarkers and subjective responses. Cancer Epidemiol Biomarkers Prev. 2013 Mar;22(3):382-9. doi: 10.1158/1055-9965.EPI-12-1097. Epub 2013 Jan 18. PMID 23334588

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the local Philadelphia area via newspaper and internet advertising. Former study participants who had agreed to be contacted for future studies were also contacted. Recruitment began October 2010 and was completed November 2011.
Pre-assignment Details: Subjects were required to complete a 5 day baseline assessment of smoking their own brand cigarette. Participants who did this were given study cigarettes. 87 participants signed consents at the first session, 3 did not finish the session. 60 subjects did the 5 day baseline smoking, returned on Day 5, were randomized and included for analysis.
Groups:
- Control: Control group: continued to smoke same, own brand cigarette.
- Experimental: Menthol to non-menthol : Switch from smoking menthol to non-menthol cigarettes.
Period: Overall Study
Arm/Group | Control | Experimental
Started | 15 | 45
Completed Period 1 Own Menthol | 15 | 45
Completed Period 2 Own or CCrush Menthol | 10 | 30
CompletedPer 3 Own or CCrush Non-menthol | 10 | 22
Completed | 10 | 22
Not Completed | 5 | 23
Not completed — Lost to Follow-up | 4 | 21
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Experimental: Group switched from menthol cigarette to non-menthol cigarette
- Control: Participants smoked their own menthol brand cigarette throughout the study.
- Total: Total of all reporting groups
Arm/Group | Experimental | Control | Total
Number analyzed (Participants) | 45 | 15 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 15 | 60
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.13 (10.9) | 37.93 (12.1) | 37.4 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 11 | 36
  Male | 20 | 4 | 24
Region of Enrollment [Number; unit: participants]
  United States | 45 | 15 | 60

OUTCOME MEASURES:

1. Primary Outcome: Smoking Topography- Puff Volume
Description: The total puff volume for a single subject is the sum of puff volumes for a subject's cigarette smoked during the study session. The mean puff volume for the subjects will be used to examine the effect of cigarette menthol on smoking topography. The values provided are the average of subjects at study Day 5 (completion of baseline smoking own cigarettes), Day 20 and Day 35.
Time Frame: over 35 day study period
Population: Those completing Study session 2 at Day 5.
Measure: Mean (Standard Error); unit: mL
Groups:
- Experimental: Experimental group switched from menthol cigarette to non-menthol cigarette
- Control: Control group smoked their own brand cigarette for entire duration of study.
Arm/Group | Experimental | Control
Number analyzed (Participants) | 45 | 15
mL
  Period 1 Own cigarette | 518 (37) | 661 (36)
  Period 2 Own cigarette or CCrush menthol | 650 (48) | 620 (41)
  Period 3 Own cigarette or CCrush non-menthol | 678 (57) | 645 (37)

2. Primary Outcome: Smoking Topography- Carbon Monoxide Boost
Description: Carbon monoxide content in exhaled breath samples is measured before and after each cigarette smoked during study sessions. CO boost is the amount in parts per million that the subject's CO increases.
Time Frame: Measured before and after each cigarette smoked at study sessions
Measure: Mean (Standard Error); unit: parts per million
Arm/Group | Experimental | Control
Number analyzed (Participants) | 45 | 15
parts per million
  Period 1 Baseline Own cigarette | 5.9 (0.8) | 5.3 (0.7)
  Period 2 Own cigarette or CCrush menthol | 3.7 (0.5) | 5.7 (0.6)
  Period 3 Own cigarette or CCrush non-menthol | 3.9 (0.5) | 5.5 (0.8)

3. Primary Outcome: Nicotine Levels
Description: Urine nicotine levels will be measured to examine the effect of cigarette menthol on harm exposure measures. Participants provided samples on the final day of each period. NNK and 1-hop were not analyzed, total nicotine metabolites were assayed.
Time Frame: 35 days
Population: Those completing Day 5, returning sample for assay
Measure: Mean (Standard Error); unit: micrograms/mL
Arm/Group | Control | Experimental
Number analyzed (Participants) | 15 | 45
micrograms/mL
  Period 1 Baseline Own cigarette | 2.2 (0.82) | 1.7 (0.3)
  Period 2 Own cigarette or CCrush non-menthol | 3.4 (1.0) | 2.7 (0.54)
  Period 3 Own cigarette or CCrush non-menthol | 2.8 (1.1) | 2.49 (.43)

4. Primary Outcome: Subjective Rating of Cigarettes
Description: Subjects completed a visual analog scale rating each cigarette smoked at each session. Subjects rated characteristics of the cigarette on a scale represented as a continuous horizontal line 10 cm long. Subjects drew an intersecting line to represent their rating. The rating reported is for the taste of the cigarette at the end of the period averaged across subjects in the group. A rating of 0 corresponds to Very Bad and a rating of 100 to Very Good for taste. There is no better or worse outcome for higher or lower ratings for taste.
Time Frame: Immediately after a cigarette smoked at the study session
Population: Completed measure
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Control | Experimental
Number analyzed (Participants) | 15 | 45
units on a scale
  Period 1 Own cigarette | 80 (8.1) | 61 (5.3)
  Period 2 Own cigarette or CCrush menthol | 72 (7.3) | 52 (5.8)
  Period 3 Own cigarette or CCrush non-menthol | 71 (6.2) | 39 (5.7)

ADVERSE EVENTS:
Description: Because this was a cigarette brand switching study there was no systematic assessment tool.
  Participants were asked about withdrawal symptoms due to the possibility of not smoking as many cigarettes.
Arm/Group | Control | Experimental
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/45
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
Attrition rate over 35 day protocol of brand switching cigarette.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No